CLINICAL TRIAL: NCT02949375
Title: A Double-blind, Randomized, Placebo-Controlled Phase 2a Trial of GRI-0621 in Patients With Chronic Liver Disease
Brief Title: Trial to Examine the Effect of Two Doses of GRI-0621 in Patients With Chronic Liver Disease
Acronym: GRI-201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative decision
Sponsor: GRI Bio Operations, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: GRI-0621-201
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Arm (Placebo Comparator): Gel capsule containing Placebo to be taken once per day
  Interventions: Drug: Placebo Comparator
- 4.5mg GRI-0621 (Active Comparator): 4.5mg GRI-0621 gel capsule to be taken once per day
  Interventions: Drug: Active Comparator:4.5mg GRI-0621
- 6mg GRI-0621 (Active Comparator): 6mg GRI-0621 gel capsule to be taken once per day
  Interventions: Drug: Active Comparator: 6.0mg GRI-0621

INTERVENTIONS:
Drug: Placebo Comparator — Placebo gel capsule to be taken daily for 28 days
  Arms: Placebo Arm
Drug: Active Comparator:4.5mg GRI-0621 — 4.5mg GRI-0621 gel capsule to be taken daily for 28 days
  Arms: 4.5mg GRI-0621
Drug: Active Comparator: 6.0mg GRI-0621 — 6.0mg GRI-0621 gel capsule to be taken daily for 28 days
  Arms: 6mg GRI-0621

SUMMARY:
Primary objectives:

To evaluate the change in serum alanine transaminase [ALT] levels from Day 0 to Day 28, following daily doses of 4.5 or 6mg of GRI-0621 compared to placebo, in patients with chronic liver disease and elevated serum levels of ALT. Serum ALT level will be used as a marker of liver inflammation.

To assess the safety and tolerability of GRI-0621 at these two doses.

Secondary objectives:

To assess the change in serum aspartate transaminase [AST] levels from baseline to Day 28, following daily doses of 4.5 or 6mg of GRI-0621 or matching placebo, in patients with chronic liver disease and elevated serum levels of AST. Serum AST level will be used as a second marker of liver inflammation.

To evaluate the response to 4.5mg GRI-0621 versus 6mg GRI-0621 in terms of the change in serum ALT levels from baseline measured at the different trial time points.

To assess changes in serum cytokeratin 18 [CK-18] levels from baseline to Day 28, following daily doses of 4.5 or 6mg of GRI-0621 or matching placebo, in patients with chronic liver disease. Serum CK-18 is used as a marker of hepatocyte cell death due to either necrosis or apoptosis.

To measure Natural Killer T lymphocyte [NKT] cell activity at baseline and at Day 28 following daily doses of 4.5 or 6mg of GRI-0621 or matching placebo.

To describe the steady-state pharmacokinetics [PK] of GRI-0621 in patients with chronic liver disease.

Exploratory objectives:

To assess the effect, if any, that the investigational product may have on serum triglyceride levels.

DETAILED DESCRIPTION:
This is a multi- centre, double-blind, randomized, placebo-controlled phase 2a trial in participants aged 18 to 65 years with chronic liver disease. It is designed to assess the safety, tolerability and efficacy of both 4.5mg and 6mg of GRI-0621 when administered once daily for 28 days.

A total of 60 participants will be randomised to received 4.5mg or 6mg of GRI-0621 or matching placebo in a 1:1:1 ratio. The investigational product will be administered orally once daily in the morning for a duration of 28 days. Participants will return to the clinic for follow-up safety and efficacy assessments on Days 7, 14, 21 and 28. Additionally, PK sampling will be performed on Days 7 and 28, and samples for immunological assays to assess the activity of NKT cells will be drawn on Days 0 (baseline) and 28. An end-of-trial follow-up visit will be performed 14 days after the last dose of the investigational product on Day 42.

The primary efficacy objective will be measured by the change from baseline to Day 28 in serum ALT levels. The baseline ALT level will be calculated as the mean of the Day -7 to -1 and Day 0 serum ALT results.

Safety and tolerability will be measured by the incidence and severity of adverse events and changes in physical examination findings, physical measurements, vital signs, ECG findings and standard laboratory safety parameters (including hematology, clinical chemistry, coagulation parameters and urinalysis).

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for participation in the trial if all of the following inclusion criteria are met:

1. Completion of the written informed consent process for trial participation prior to all trial-related procedures, including HIV testing.
2. Male or female participants aged 18 to 65 years.
3. Female participants of child-bearing potential must practice an effective method of birth control from four weeks prior to randomization and agree to continue this until 6 months after the completion of the end-of-trial follow-up visit. Effective birth control must include two methods, one of which must be a barrier method. Female participants are considered not to be of child-bearing potential if they are post-menopausal (12 months of spontaneous amenorrhoea with an appropriate clinical profile, or 6 months of spontaneous amenorrhoea with local laboratory serum follicle-stimulating hormone [FSH] levels in keeping with post-menopause) or surgically sterile (after bilateral oophorectomy, hysterectomy or salpingectomy). For the purpose of this trial any participant who has had a tubal ligation will not be considered surgically sterile due to the teratogenic nature of this class of chemical entities.
4. Female participants of child-bearing potential must have negative serum and urine pregnancy tests at screening and randomization respectively.
5. History of chronic liver disease [CLD] as a result of viral hepatitis, alcoholic steatohepatitis [ASH] or non-alcoholic steatohepatitis [NASH].
6. Evidence of viral hepatitis, ASH or NASH as described beneath:

   * Viral Hepatitis:

     * Hepatitis C virus [HCV] infection as confirmed by the presence of HCV RNA (determined by PCR) and no other cause of liver disease or
     * Hepatitis B virus [HBV] infection as confirmed by the presence of HBV DNA > 104 copies/ml (determined by the Roche COBA TaqMan HBV DNA assay) and no other cause for liver disease or
     * Hepatitis C and B co-infection (as defined above) OR
   * ASH:

     * Findings and history consistent with the diagnosis of ASH in the opinion of the investigator OR
   * NASH:

     * Absence of viral hepatitis and
     * A history of no or minimal alcohol use and
     * Findings and history consistent with the diagnosis of NASH in the opinion of the investigator
7. Body Mass Index (BMI) of 18 to 39kg/m2.
8. Weight ≥ 45kg
9. ALT > 1.5 x ULN but less than 10 x ULN on two occasions during the screening period (Day -28 to Day -1). The second occasion must be between Day -7 and Day -1.
10. An ability to communicate well with the investigator and to understand and comply with the requirements of the trial.
11. Agree to stay in contact with the trial site for the duration of the trial, provide updated contact information as necessary.

Exclusion Criteria:

A participant will not be eligible for trial participation if any of the following exclusion criteria are met:

1. Use of any other investigational drug within 30 days or five half-lives (whichever is longer) of the first dose of GRI-0621.
2. Current pregnancy or lactation.
3. A history of anaphylaxis or severe hypersensitivity to any drugs.
4. A known hypersensitivity to any component of the investigational product or to any other retinoids.
5. ALT or AST > 10 x ULN on any occasion during the screening period (Day -28 to Day -1)
6. ALT or AST known to have been > 10 X ULN on any occasion during the 2 months prior to screening.
7. Any of the following laboratory abnormalities at screening:

   * Serum creatinine > 1.5 x ULN
   * Hemoglobin < 10.0 g/L
   * Platelets < 75 x 109/L
   * White cell count < 3.0 x 109/L.
8. Known hypothyroidism requiring treatment or laboratory results suggestive of hypothyroidism at screening (thyroxine [T4] < LLN and thyroid-stimulating hormone [TSH] > ULN).
9. Any clinically significant ECG abnormalities.
10. Current or recent (during the 3 months prior to screening) or required treatment for tuberculosis infection.
11. A history of any malignancy (other than treated localized basal cell carcinoma of the skin) in the last 5 years.
12. A history or known presence of osteoporosis.
13. A history of arthritic conditions requiring treatment with symptom- or disease-modifying drugs for > 4 weeks.
14. A history of atopic dermatitis.
15. History or presence of decompensated liver disease
16. Previous histological evidence of hepatic fibrosis stage > 3.
17. The presence of any acute disorder that could further compromise the hepato-biliary system including but not limited to acute infectious or alcoholic hepatitis, acute pancreatitis, biliary obstruction and cholecystitis.
18. History or presence of hepatocellular carcinoma, hepatic abscess, biliary obstruction or portal vein thrombosis as confirmed by ultrasound, CT or MRI scans.
19. A history of severe gastro-intestinal bleeding requiring blood transfusion therapy (packed cells or whole blood).
20. Any surgical or medical condition other than CLD which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the participant or the objectives of the trial including but not limited to inflammatory bowel disease, major gastro-intestinal surgery (e.g. gastrectomy, gastroenterostomy or bowel resection) or pancreatic injury.
21. A history of hemachromatosis, Wilson's disease, alpha-1-antitrypsin deficiency or celiac disease.
22. Previous organ or hematopoietic transplantation.
23. HIV infection confirmed by a positive HIV test result.
24. Any other medical condition which, in the opinion of the investigator, could affect the participant's health during trial participation or could compromise his/her ability to participate in the trial. This includes but is not limited to significant cardiovascular, respiratory, renal, neurological, hematological, immunological, endocrinological or metabolic disorders.
25. Any psychiatric or mental disorder which could limit the validity of the informed consent or the participant's ability to comply with the protocol requirements.
26. A history of drug abuse during the 12 months prior to screening, or evidence of such abuse as indicated by urine testing for drugs of abuse at screening that, in the opinion of the investigator, may be indicative of potential participant adherence issues during the course of the trial.
27. In the opinion of the investigator, the participant is not reliable to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in serum ALT levels from Day 0 (baseline) to Day 28 | 0 and 28 days
  To evaluate the change in serum ALT levels from baseline to Day 28, following daily doses of 4.5 or 6mg of GRI-0621 compared to placebo, in patients with chronic liver disease and elevated serum levels of ALT. Serum ALT level will be used as a marker of liver inflammation.

SECONDARY OUTCOMES:
Change in serum AST levels from Day 0 (baseline) to Day 28 | 0 and 28 days
  To assess the change in serum AST levels from baseline to Day 28, following daily doses of 4.5 or 6mg of GRI-0621 or matching placebo, in patients with chronic liver disease and elevated serum levels of AST. Serum AST level will be used as a second marker of liver inflammation.
Response to 4.5mg GRI-0621 versus 6mg GRI-0621 in terms of the change in serum ALT levels from Day 0 (baseline) measured at the different trial time points. | 0 and 28 days
Changes in serum cytokeratin 18 (CK-18) levels from Day 0 (baseline) to Day 28, | 0 and 28 days
  To assess changes in serum cytokeratin 18 (CK-18) levels from Day 0 to Day 28, following daily doses of 4.5 or 6mg of GRI-0621 or matching placebo, in patients with chronic liver disease. Serum CK-18 is used as a marker of hepatocyte cell death due to either necrosis or apoptosis.
NKT cell activity measured by multi-color flow cytometry at Day 0 (baseline) and at Day 28 following daily doses of 4.5 or 6mg of GRI-0621 or matching placebo. | 0 and 28 days
Measurement of GRI-0621 peak plasma concentration [Cmax] on Day 7 and Day 28. | 7 and 28 days
Measurement of GRI-0621 time to reach Cmax [Tmax]. | 7 and 28 days
Measurement of GRI-0621 half life [t1/2] | 7 and 28 days
Measurement of GRI-0621 clearance [CL] on Days 7 and 28 | 7 and 28 days
Measurement of GRI-0621 volume of distribution [Vd] on Days 7 and 28 | 7 and 28 days

OTHER OUTCOMES:
Effect, if any, that the investigational product may have on serum triglyceride levels. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mpho K Kgomo, MBBCH, Principal Investigator — Department Head; Gastroenetrology
Locations (1):
- Steve Biko Academic Hospital, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No